CLINICAL TRIAL: NCT03420417
Title: Study of the Respiratory Mechanics Characteristics With Esophageal PREssure Measurements in Mechanically Ventilated Patients in IntensivE caRe Unit
Brief Title: Respiratory Mechanics in Intensive Care Patients
Acronym: PREMIER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 49RC17_0200
Record Dates: First submitted 2018-01-18; First posted 2018-02-05 (Actual); Last update posted 2018-03-30 (Actual); Status verified 2018-02

CONDITIONS: Intensive Care; Ventilator Lung
Keywords: Mechanical ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assessement of respiratory mechanics (Experimental): Measurement of respiratory mechanics characteristics
  Interventions: Device: Esophageal pressure measurement

INTERVENTIONS:
Device: Esophageal pressure measurement — Use of a nasogastric tube equipped with esophageal balloon to assess respiratory mechanics

SUMMARY:
This study aims at assessing the respiratory mechanics of intubated patients in intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 18 years
* Invasive mechanical ventilation on tracheal tube
* Treatment with neuromuscular blocking agents
* Nasogastric tube needed for enteral nutrition

Exclusion Criteria:

* Lack of free and informed consent
* Pregnant or breastfeeding woman
* Contra-indication to esophageal pressure measurement catheter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-03-28 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Chest wall compliance measurement (mL/cmH2O) | 1 hour

SECONDARY OUTCOMES:
lung compliance measurement (mL/cmH2O) | 1 hour
End expiratory lung volume (mL) | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: François Beloncle, MCU-PH, Principal Investigator — University Hospital, Angers
Locations (1):
- University hospital, Angers, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beloncle FM, Richard JC, Merdji H, Desprez C, Pavlovsky B, Yvin E, Piquilloud L, Olivier PY, Chean D, Studer A, Courtais A, Campfort M, Rahmani H, Lesimple A, Meziani F, Mercat A. Advanced respiratory mechanics assessment in mechanically ventilated obese and non-obese patients with or without acute respiratory distress syndrome. Crit Care. 2023 Sep 4;27(1):343. doi: 10.1186/s13054-023-04623-2. PMID 37667379
- [Derived] Beloncle FM, Merdji H, Lesimple A, Pavlovsky B, Yvin E, Savary D, Mercat A, Meziani F, Richard JC. Gas Exchange and Respiratory Mechanics after a Cardiac Arrest: A Clinical Description of Cardiopulmonary Resuscitation-associated Lung Edema. Am J Respir Crit Care Med. 2022 Sep 1;206(5):637-640. doi: 10.1164/rccm.202111-2644LE. No abstract available. PMID 35579690